CLINICAL TRIAL: NCT03560518
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of Rapastinel as Monotherapy in Patients With Major Depressive Disorder
Brief Title: Study of Rapastinel as Monotherapy in Patients With MDD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision to stop the program.
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAP-MD-32
Record Dates: First submitted 2018-06-07; First posted 2018-06-18 (Actual); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Depressive Disorder, Major
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — GLYX-13 peptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rapastinel 450mg (Experimental): Rapastinel 450 mg (prefilled syringe, weekly intravenous IV administration)
  Interventions: Drug: Rapastinel
- Rapastinel 900mg (Experimental): Rapastinel 900 mg (prefilled syringe, weekly intravenous IV administration)
  Interventions: Drug: Rapastinel
- Placebo (Placebo Comparator): Placebo (prefilled syringe, weekly IV administration)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapastinel — Rapastinel (prefilled syringe, weekly intravenous IV administration)
  Arms: Rapastinel 450mg; Rapastinel 900mg
Drug: Placebo — Placebo (prefilled syringe, weekly IV administration)
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy, safety, and tolerability of 450 milligrams (mg) and 900 milligrams (mg) of Rapastinel, compared to placebo in participants with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for MDD
* Current major depressive episode of at least 8 weeks and not exceeding 18 months in duration at Visit 1
* Treatment naive in the current episode or have inadequate response to 1-3 antidepressant therapies given at adequate dose and duration in the current episode
* If female of childbearing potential, have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test

Exclusion Criteria:

* DSM-5-based diagnosis of any disorder other than MDD that was the primary focus of treatment within 6 months before Visit 1
* Lifetime history of meeting DSM-5 criteria for:
* Schizophrenia spectrum or other psychotic disorder
* Bipolar or related disorder
* Major neurocognitive disorder
* Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study
* Dissociative disorder
* Posttraumatic stress disorder
* MDD with psychotic features
* Significant suicide risk, as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hoogerheyde, Study Director — Allergan
Locations (40):
- United States (40):
  - Alea Research, Phoenix, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - California Pharmaceutical Research Institute, Inc., Anaheim, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - Synergy Research San Diego, National City, California
  - Excell Research Inc., Oceanside, California
  - NRC Research Institute, Orange, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Neuroscience Research Medical Group,Inc., Sherman Oaks, California
  - Viking Clinical Research Ltd., Temecula, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Research Centers of America, LLC, Hollywood, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Innova Clinical Trials, Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Institute for Advanced Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Iris Research, Inc., Smyrna, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Pharmasite Research, Inc., Baltimore, Maryland
  - CBH Health, LLC, Gaithersburg, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Bioscience Research LLC, Mount Kisco, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - New Hope Clinical Research Inc., Charlotte, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - Donald J. Garcia, Jr., MD, PA, Austin, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Period: Double Blind Treatment Period
Arm/Group | Placebo | Rapastinel 450mg | Rapastinel 900mg
Started | 147 | 145 | 147
Completed | 122 | 116 | 124
Not Completed | 25 | 29 | 23
Not completed — Miscellaneous Reasons | 1 | 0 | 0
Not completed — Study Terminated by the Sponsor | 6 | 9 | 10
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Pregnancy | 0 | 2 | 0
Not completed — Lost to Follow-up | 5 | 6 | 6
Not completed — Withdrawal by Subject | 10 | 6 | 5
Not completed — Lack of Efficacy | 2 | 1 | 1
Not completed — Adverse Event | 0 | 3 | 1
Period: Safety Follow-Up Period
Arm/Group | Placebo | Rapastinel 450mg | Rapastinel 900mg
Started | 10 | 17 | 22
Completed | 10 | 17 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The modified Intent-to-Treat (mITT) Population will consist of all patients in the Safety Population who had at least 1 postbaseline assessment of the MADRS total score or S-STS total score.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rapastinel 450mg | Rapastinel 900mg | Total
Number analyzed (Participants) | 146 | 144 | 147 | 437
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (14.35) | 45.8 (14.02) | 44.5 (13.14) | 44.7 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 100 | 101 | 299
  Male | 48 | 44 | 46 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 30 | 21 | 76
  Not Hispanic or Latino | 121 | 114 | 126 | 361
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 1 | 6
  Asian | 4 | 1 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2 | 4
  Black or African American | 31 | 27 | 35 | 93
  White | 106 | 111 | 103 | 320
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 86.42 (18.11) | 88.20 (18.61) | 85.33 (20.71) | 86.64 (19.18)
Height [Mean (Standard Deviation); unit: cm] | 168.41 (9.66) | 168.75 (9.83) | 168.57 (10.21) | 168.58 (9.88)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.54 (6.39) | 30.96 (6.13) | 30.00 (6.96) | 30.50 (6.50)
Montgomery-Asberg Depression Rating Scale (MADRS) total score at baseline [Mean (Standard Deviation); unit: Score on a Scale] — The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression.
  Score on a Scale | 35.4 (4.50) | 35.1 (4.71) | 35.9 (4.69) | 35.5 (4.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at End of Treatment (End of Week 6)
Description: The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
Time Frame: Baseline to end of Week 6
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Rapastinel 450mg | Rapastinel 900mg
Number analyzed (Participants) | 146 | 144 | 147
Scores on a scale | -13.8 (11.93) | -13.2 (11.62) | -11.3 (11.36)

2. Secondary Outcome: Change From Baseline in MADRS Total Score at Day 1 Post-first Dose of Treatment
Description: as for outcome 1
Time Frame: Baseline to Day 1 post-first dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Rapastinel 450mg | Rapastinel 900mg
Number analyzed (Participants) | 146 | 144 | 147
Scores on a Scale | -11.0 (9.47) | -9.0 (9.18) | -8.3 (8.36)

ADVERSE EVENTS:
Time Frame: The study consisted of a 6 week double-blind treatment period, followed by a 2-week safety follow-up period.
Description: The Safety Population consists of all randomized patients who received at least 1 dose of randomized IP.
Arm/Group | Placebo | Rapastinel 450mg | Rapastinel 900mg
All-Cause Mortality (participants affected / at risk) | 0/147 | 1/145 | 0/147
Serious Adverse Events (participants affected / at risk) | 2/147 | 2/145 | 1/147
Other Adverse Events (participants affected / at risk) | 15/147 | 28/145 | 21/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | Rapastinel 450mg (N=145) | Rapastinel 900mg (N=147)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | Rapastinel 450mg (N=145) | Rapastinel 900mg (N=147)
Headache (Nervous system disorders) | 11 | 13 | 11
Nasopharyngitis (Infections and infestations) | 6 | 9 | 8
Dysgeusia (Nervous system disorders) | 0 | 11 | 4

LIMITATIONS AND CAVEATS:
Due to study termination, the target number of participants needed to achieve target power and statistically reliable results was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT03560518/SAP_000.pdf
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT03560518/Prot_001.pdf